CLINICAL TRIAL: NCT00073346
Title: Cognitive and Behavioral Treatment of Compulsive Hoarding
Brief Title: Pilot Trial of Cognitive and Behavioral Treatment of Compulsive Hoarding Compared to Wait List Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH068539 (NIH); R21MH068539 (NIH); DATR A2-AIA
Record Dates: First submitted 2003-11-19; First posted 2003-11-21 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Hoarding Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Hoarding Disorder

STUDY DESIGN:
Intervention Model Description: active treatment versus wait list control
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive behavior therapy for hoarding disorder (Experimental): Cognitive behavior therapy included 26 sessions of motivational enhancements; skills training for sorting, organizing and problem solving; direct practice not acquiring new items and discarding possessions to remove clutter and organize possessions; cognitive therapy to evaluate beliefs about possessions; and relapse prevention skills.
  Interventions: Behavioral: Cognitive Behavioral Treatment
- Wait list control (No Intervention): Participants waited to receive treatment for 12 weeks

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment
  Arms: cognitive behavior therapy for hoarding disorder

SUMMARY:
This study developed and tested a specialized cognitive and behavioral treatment for the symptoms of hoarding disorder, including excessive acquiring, difficulty discarding items, and extensive clutter in the home.

DETAILED DESCRIPTION:
Compulsive hoarding is characterized by excessive acquisition of possessions, difficulty discarding possessions, and excessive clutter. This condition is resistant to standard pharmacological and psychotherapeutic interventions that have proven effective in treating other obsessive compulsive spectrum disorders. This study aimed to determine the effectiveness of a specialized cognitive behavioral therapy (CBT) designed for treating hoarding symptoms.

This study consists of three phases. In Phase 1, pilot data from previous studies were examined to develop an intervention suitable for use in a waitlist trial. In Phase 2, pilot study information were used to develop and test a treatment manual for compulsive hoarding. During this phase, treatment was applied flexibly to allow for variations in treatment duration and choice of techniques. During Phase 3, participants were randomly assigned to 26 weekly sessions of CBT or to a 12-week wait-list control, followed by active treatment for a fixed duration of 26 sessions. Therapist adherence and competence were assessed through audiotaped therapy sessions.

ELIGIBILITY:
Inclusion criteria:

* Display at least moderately severe hoarding symptoms
* Must live within 45 minutes of Boston, MA or Hartford, CT

Exclusion criteria:

* Ten or more sessions of cognitive behavior therapy for hoarding
* Concurrent psychotherapy or medications
* Suicidal, psychotic, or other psychiatric symptoms requiring hospitalization
* Compulsive buying symptoms that are part of a manic phase of bipolar disorder
* Mental retardation, dementia, brain damage, or other cognitive dysfunction that would interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-09-01 (Actual); Primary Completion 2006-12-01 (Actual); Study Completion 2008-07-09 (Actual)

PRIMARY OUTCOMES:
Saving Inventory-Revised | change from baseline to week 12; change from baseline to week 26
  Self-report questionnaire of hoarding severity; total score range = 0 to 92; higher values indicate more symptoms

SECONDARY OUTCOMES:
Hoarding Rating Scale | change from baseline to week 12; change from baseline to week 26
  Interviewer measure with 5 questions to assess hoarding severity; total score range = 0 to 40; higher values indicate more symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Gail Steketee, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Hartford Hospital, Institute of Living, Hartford, Connecticut
  - BostonUCRC, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
De-identified data have been shared with investigators working on hoarding relevant projects such as assessment of hoarding and meta-analyses of treatment outcome for hoarding disorder. Sharing of de-identified data will be considered upon request.

REFERENCES:
- See also: Click here for more information about compulsive hoarding. — http://www.ocfoundation.org